CLINICAL TRIAL: NCT01633528
Title: To Evaluate the Effect of Low Dose Aspirin in Increasing the Chance of Pregnancy in Frozen Embryo Transfer Cycles
Brief Title: The Effect of Low Dose Aspirin in Increasing the Chance of Pregnancy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Royan-Emb-014
Record Dates: First submitted 2012-05-14; First posted 2012-07-04 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2012-03

CONDITIONS: Infertility
Keywords: low dose aspirin endometrial thickness pregnancy rate ICSI IVF embryo transfer
MeSH Terms: conditions — Infertility | interventions — acetylsalicylic acid lysinate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Asprin (Experimental): With the onset of endometrial preparation and estrogen treatment, the study group will receive 100 mg of oral aspirin.
  Interventions: Drug: Asprin
- placebo (Placebo Comparator): With the onset of endometrial preparation and estrogen treatment, the control group will receive placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Asprin — 100 mg
  Arms: Asprin
Drug: placebo — 100mg
  Arms: placebo

SUMMARY:
It has been reported that low-dose aspirin and Heparin would lead to an increased Pregnancy rate in patients undergoing IVF-ET. Low-dose aspirin may improve uterine and ovarian perfusion and that aspirin might enhance endometrial receptivity and ovarian responsiveness as well, which could result in better implantation and pregnancy rates after IVF or ICSI treatment. This study assesses potential effects of low-dose aspirin (100 mg daily) on pregnancy rate following frozen embryo transfer.

DETAILED DESCRIPTION:
In the present randomized double-blind prospective study, the patients will be randomly assigned to the study and control groups. With the onset of endometrial preparation and estrogen treatment, the study group will receive 100 mg of oral aspirin and the control group will be given placebo. When endometrial thickness will be found between 8-14 mm, therapy with progesterone (100 mg IM daily) will be started and embryo transfer will be performed 48 to 72 hours later. Doppler ultrasonography also is done to calculate Resistive Index (RI) and Pulsatility Index (PI), the day after progesterone administration.

βHCG will be assessed 14 days after ET. If a pregnancy will be achieved, the patients in study and control groups will be instructed to continue the aspirin or placebo through 5 weeks and if the pregnancy test result will be negative, the treatment with aspirin or placebo will be stopped. The patients will be followed until 20 weeks of gestation and the results of treatment cycle will be compared in two groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients with "long or antagonist" protocol
* Women who did not achieve a pregnancy following a fresh embryo transfer or women whom their embryos had not been transferred due to OHSS
* The women who had frozen embryos available for another transfer no contraindications for aspirin

Exclusion Criteria:

* The patients with history of recurrent abortion

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2012-05; Primary Completion 2012-09 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Pregnancy rate | 6 weeks
  evaluation the clinical pregnancy rate 6 weeks after emberyo transfering.

SECONDARY OUTCOMES:
Implantation rate | 8 weeks
  Evaluation the implantation rate after emberyo transfer in women who use low dose of aspirin
Miscarriage rate | 12 weeks
  Evaluation the miscariage rate after emberyo transfer in women who use asprin.

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Gourabi, PhD, Study Chair — Head of Royan institute; Tahereh Madani, MD, Study Director — Endocrinology and Female Infertility Department; Firoozeh Ahmadi, MD, Principal Investigator — Reproductive Imaging Department; Poopak Eftekhary, PhD, Principal Investigator — Embryology Department
Locations (1):
- Royan Institute, Tehran, Iran

REFERENCES:
- See also: Related Info — http://Royaninstitute.org